CLINICAL TRIAL: NCT04330079
Title: Effects of dapaglifloziN Therapy on Myocardial Perfusion Reserve in Prediabetic Patients With Stable coronarY Artery Disease (ENTRY Trial)
Brief Title: Effects of dapaglifloziN Therapy on Myocardial Perfusion Reserve in Prediabetic Patients With Stable coronarY Artery Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment. (Difficulty in selecting subjects)
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENTRY trial
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease; Prediabetic State
Keywords: Dapagliflozin; Lifestyle modification; Myocardial perfusion reserve
MeSH Terms: conditions — Coronary Artery Disease; Prediabetic State | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin 10mg
- Lifestyle modification (Other)
  Interventions: Other: Lifestyle modification

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10mg once daily for 6 months.
  Arms: Dapagliflozin
Other: Lifestyle modification — lifestyle modification (diet and exercise) for 6 months
  Arms: Lifestyle modification

SUMMARY:
The purpose of this study is to investigate the effects of dapagliflozin therapy on myocardial perfusion reserve (MPR) using dynamic SPECT examination in prediabetic patients with stable CAD.

Dapagliflozin therapy versus lifestyle modification improves myocardial perfusion reserve in prediabetic patients with stable CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age
2. Prediabetes by ADA criteria (fasting glucose 100-125mg/dl, or HbA1C 5.7-6.4%)
3. Stable coronary artery disease
4. Global myocardial perfusion reserve (MPR) index < 2.0
5. The patient or guardian agrees to the study protocol and the schedule of clinical and dynamic SPECT follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Contraindications to dapagliflozin
2. Significant renal disease manifested by eGFR<30 ml/min/1.73m²
3. Unstable or rapidly progressing renal disease
4. Acute coronary syndrome, or any other major cardiovascular events within the previous 6 months
5. Stent placement, or coronary artery bypass graft surgery within the previous 6 months
6. Planned revascularization within 6 months
7. Significant disease (diameter stenosis >70% by coronary CT angiography) in major epicardial coronary arteries
8. Heart failure requiring loop diuretics
9. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
10. Contraindication to adenosine stress test
11. Current treatment for the active cancer
12. Women of child bearing potential who are not willing to use a medically accepted method of contraception. Patient's pregnancy confirmed by positive pregnancy test, or breast-feeding.
13. Expected life expectancy < 1 year
14. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests which, in the judgment of the investigator, would preclude safe completion of the study.
15. Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Percent change in global myocardial perfusion reserve (MPR) index | 6months

SECONDARY OUTCOMES:
Percent change in regional myocardial perfusion reserve (MPR) index | 6months
absolute changes in global MPR index | 6months
absolute changes in regional MPR index | 6months
Change in body weight | 6months
Change in blood pressure(systolic, diastolic both ) | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Whan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided